CLINICAL TRIAL: NCT03197090
Title: Handheld ECG Tracking of In-hOspital Atrial Fibrillation - The HECTO-AF Trial
Brief Title: Handheld ECG Tracking of In-hOspital Atrial Fibrillation
Acronym: HECTO-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor patient recruitment and limited resources
Sponsor: Stéphane Cook, Prof (Other)
Responsible Party: Sponsor-Investigator, Stéphane Cook, Prof, Sponsor-Investigator, University of Freiburg
Organization: University of Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HECTO-AF Trial
Record Dates: First submitted 2017-06-10; First posted 2017-06-23 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: Screening; Zenicor
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zenicor ON (Experimental): Patients allocated to the experimental group will undergo systematic short ECG monitoring
  Interventions: Device: Zenicor ECG
- Zenicor OFF (No Intervention): In patients allocated to the control group, usual diagnostic procedures for detection of atrial fibrillation will be employed according to ESC Guidlines.

INTERVENTIONS:
Device: Zenicor ECG — Participants will place their thumbs on the device twice daily and whenever they notice palpitations.
  Arms: Zenicor ON

SUMMARY:
This is a single center, open label, randomized control trial to assess the efficacy of a one-lead ECG handheld device (Zenicor) for the detection of previously unknown atrial fibrillation (AF) in hospitalized patients.

All patients admitted to the internal medicine department of the Hospital Fribourg throughout the study period will be screened for study enrollment. Patients < 18 years, with known or previously documented atrial fibrillation, patients with a cardiac pacemaker, and implantable cardioverter-defibrillator or intra-cardiac monitoring device will be excluded from the present trial. The study population will consist of approximately 800 patients in each group at the University of Fribourg Medical Center. Patients must meet all eligibility criteria for inclusion into the study.

Patients allocated to the treatment group will undergo twice daily monitoring with the handheld Zenicor ECG. Additional recordings will be obtained whenever patients notice palpitations. Recordings will be obtained in the presence of specially trained nurses. The recordings will then be validated through a web-based interface offered by Zenicor. The one-lead ECGs will be reviewed by the investigating physicians through the Web-based analysis service (Zenicor-ECG Doctor System) to assess the presence of atrial fibrillation.

The primary end point of the study is the percentage of newly detected atrial fibrillation at 6 months

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the internal medicine department of the University and Hospital Fribourg throughout the study period will be screened for study enrollment.

Exclusion Criteria:

* Patients with known or previously documented atrial fibrillation, patients with a cardiac pacemaker, and implantable cardioverter-defibrillator or intra-cardiac monitoring device will be excluded from the present trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Newly detected in-hospital AF | During hospitalizaion
  Proportion of newly detected atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane P Cook, MD, Study Chair — University of Freiburg
Locations (1):
- University and hospital of Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Svennberg E, Engdahl J, Al-Khalili F, Friberg L, Frykman V, Rosenqvist M. Mass Screening for Untreated Atrial Fibrillation: The STROKESTOP Study. Circulation. 2015 Jun 23;131(25):2176-84. doi: 10.1161/CIRCULATIONAHA.114.014343. Epub 2015 Apr 24. PMID 25910800
- [Background] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Background] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Derived] Mancinetti M, Schukraft S, Faucherre Y, Cook S, Arroyo D, Puricel S. Handheld ECG Tracking of in-hOspital Atrial Fibrillation (HECTO-AF): A Randomized Controlled Trial. Front Cardiovasc Med. 2021 May 4;8:681890. doi: 10.3389/fcvm.2021.681890. eCollection 2021. PMID 34017869
- [Derived] Schukraft S, Mancinetti M, Hayoz D, Faucherre Y, Cook S, Arroyo D, Puricel S. Handheld ECG Tracking of in-hOspital Atrial Fibrillation The HECTO-AF trial Clinical Study Protocol. Trials. 2019 Jan 30;20(1):92. doi: 10.1186/s13063-019-3189-7. PMID 30700332